CLINICAL TRIAL: NCT01734070
Title: Role of Cherry Consumption in Reducing Risk Factors for Human Chronic Inflammatory Diseases
Brief Title: Role of Cherry Consumption in Reducing Risk Factors for Chronic Inflammatory Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: California Cherry Board (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FL40
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Inflammation; Cardiovascular Diseases
Keywords: anthocyanins; catechins; chlorogenic acid; flavanol glycosides
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cherry consumption (Experimental): Volunteers will supplement their diets with 280 grams/day of pitted Bing cherries by replacing an equivalent amount of carbohydrate calories. We will prefer that the subjects split the cherries into three equal portions and consume one with each meal; however, this will not be mandatory.
  Interventions: Other: Cherry consumption

INTERVENTIONS:
Other: Cherry consumption — Volunteers will eat 280 grams/day of pitted Bing cherries by replacing an equivalent amount of carbohydrate calories.

SUMMARY:
The goal of this study is to examine if chronic cherry consumption will decrease lipid peroxidation and serum concentration of inflammatory markers in human subjects with elevated serum C reactive protein (CRP), and to examine the relationship between serum concentrations of CRP and polyphenols. The investigators hypothesize that cherry consumption will reduce serum concentration of inflammatory markers, including CRP, inflammatory cytokines and adhesion molecules.

DETAILED DESCRIPTION:
The study will last a total of 64 days with three different metabolic periods. First 8 days will be period 1, when base line fasting blood samples will be collected on day 1 and 8. For the next 28 days (period 2 or intervention period) subjects will supplement their diets with 280 g/d of pitted Bing cherries by replacing an equivalent amount of carbohydrate calories. We will prefer that the subjects split the cherries into three equal portions and consume one with each meal; however, this will not be mandatory. Subjects will be asked to record all foods and drinks consumed for three 24-hr periods during the study. Fasting blood samples will be drawn on study days 22 and 36 (14 and 28 day after the start of cherry consumption). The third period of 28 days will be post-intervention, when the subjects will return to their normal diets without cherries. Post-intervention blood samples will be drawn on study day 64. All blood draws will follow a 12-hour fast. Blood samples will be processed within one hour of draw and the plasma stored frozen in different aliquots, until analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 45-65 years of age
* serum CRP concentrations between 3-25 mg/L
* BMI < 35 kg/m2

Exclusion Criteria:

* BMI > 35 kg/m2
* current infection
* taking anti-inflammatory medications

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-05; Primary Completion 2003-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Change in lipid peroxidation | baseline, day 36, and day 64
  The study will last a total of 64 days with three different metabolic periods. First 8 days will be period 1, when baseline fasting blood samples will be collected on day 1 and 8. For the next 28 days (period 2 or intervention period) subjects will supplement their diets with 280 g/d of pitted Bing cherries by replacing an equivalent amount of carbohydrate calories. Fasting blood samples will be drawn on study day 36. The third period of 28 days will be post-intervention, when the subjects will return to their normal diets without cherries. Post-intervention blood samples will be drawn on study day 64.

SECONDARY OUTCOMES:
Change in serum concentration of inflammatory markers | baseline, day 36 and day 64
  The study will last a total of 64 days with three different metabolic periods. First 8 days will be period 1, when baseline fasting blood samples will be collected on day 1 and 8. For the next 28 days (period 2 or intervention period) subjects will supplement their diets with 280 g/d of pitted Bing cherries by replacing an equivalent amount of carbohydrate calories. Fasting blood samples will be drawn on study day 36. The third period of 28 days will be post-intervention, when the subjects will return to their normal diets without cherries. Post-intervention blood samples will be drawn on study day 64.

CONTACTS AND LOCATIONS:
Overall Officials: Darshan Kelley, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Derived] Kelley DS, Adkins Y, Reddy A, Woodhouse LR, Mackey BE, Erickson KL. Sweet bing cherries lower circulating concentrations of markers for chronic inflammatory diseases in healthy humans. J Nutr. 2013 Mar;143(3):340-4. doi: 10.3945/jn.112.171371. Epub 2013 Jan 23. PMID 23343675
- See also: USDA, ARS, WHNRC — http://www.ars.usda.gov/Main/docs.htm?docid=11240